CLINICAL TRIAL: NCT00380159
Title: An Open-Label, 48-Week Extension Study of Elvucitabine Administered In Combination With Background Antiretroviral Agents in Participants Who Have Completed 14 Days of Treatment in Protocol ACH443-014A.
Brief Title: Open-Label, 48-Week Extension Study of Elvucitabine in Combination With Background Antiretroviral Therapy (ART) for Participants Who Have Completed Study ACH443-014A
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Achillion, a wholly owned subsidiary of Alexion (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACH443-018
Record Dates: First submitted 2006-09-21; First posted 2006-09-25 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Human Immunodeficiency Virus (HIV)-1 Infection
Keywords: Extension study to Study ACH443-014A
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — dexelvucitabine; Lamivudine; Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Elvucitabine — Elvucitabine 10 mg in combination with background ART
Drug: Lamivudine
Drug: Emtricitabine

SUMMARY:
To assess the safety of 48 weeks of treatment with 10 milligrams (mg) of elvucitabine in combination with background antiretroviral therapy (ART) in participants who completed Study ACH443-014A and meet the inclusion and exclusion criteria.

DETAILED DESCRIPTION:
This study is an open-label extension study for participants who have completed 14 days of treatment in Study ACH443-014A and meet all inclusion and exclusion criteria. Elvucitabine treatment (10 mg) will begin on Day 1 (Day 15 following completion of Study ACH443-014A) for all consenting participants in combination with background ART as determined by the Principal Investigator. Participants will have clinical and laboratory assessments every 2 weeks for the first 8 weeks and then every 4 weeks to Week 48.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have completed 14 days of treatment in Study ACH443-014A and who, in the Investigator's judgment, remain candidates to receive elvucitabine together with background ART.

Exclusion Criteria:

* Failure to meet inclusion criteria

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2006-09; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To Assess The Safety Of 48 Weeks Of 10 mg/daily (QD) Of Elvucitabine In Combination With ART | September 2008

SECONDARY OUTCOMES:
To Describe The Anti-viral Activity Of Elvucitabine In Combination With ART As Measured By Plasma HIV-1 Ribonucleic Acid (RNA) Over 24 Weeks | September 2008

CONTACTS AND LOCATIONS:
Locations (7):
- United States (2):
  - Clinical Trial Site, Atlanta, Georgia
  - Clinical Trial Site, Cincinnati, Ohio
- Clinical Trial Site, Santo Domingo, Dominican Republic
- Germany (3):
  - Clinical Trial Site, Berlin
  - Clinical Trial Site, Bonn
  - Clinical Trial Site, Cologne
- Clinical Trial Site, Madrid, Spain